CLINICAL TRIAL: NCT06062745
Title: A Pilot Study for Detection of PSMA-Low Castration Resistant and Neuroendocrine Prostate Cancer With 18F-fluciclovine PET/CT Imaging
Brief Title: Pilot Study for Detection of PSMA-Low CRPC-NE Tumors With Fluciclovine PET/CT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Blue Earth Diagnostics (Industry)
Responsible Party: Principal Investigator, Heather A. Jacene, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-267
Record Dates: First submitted 2023-09-13; First posted 2023-10-02 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Advanced Prostate Cancer; Metastatic Prostate Cancer; Metastatic Prostate Neuroendocrine Carcinoma
Keywords: Advanced Prostate Cancer; Metastatic Prostate Cancer; Metastatic Prostate Neuroendocrine Carcinoma; PSMA-Low Castration Resistant Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — fluciclovine F-18; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 18F-fluciclovine (Experimental): Participants with low prostate-specific membrane antigen (PSMA) expression or neuroendocrine prostate cancer will receive:
  * 18F-fluciclovine PET/CT within 6 weeks of standard of care exam and 68Ga-PSMA PET/CT
  * 2x Blood test at time of 18F-fluciclovine PET/CT and prior to treatment as determined by participants primary oncologist
  Interventions: Drug: 18F-fluciclovine; Device: PET/CT

INTERVENTIONS:
Drug: 18F-fluciclovine — 18F-fluciclovine is a radiotracer targeting amino-acid transporters.Radiotracers are compounds or drugs that are attached to small amounts of a radioactive substance to make images of processes that are happening in the body
  Other Names: Axumin
Device: PET/CT — Positron emission tomography/computed tomography (PET/CT) uses small amounts of radioactive materials called radiotracers, a special camera and a computer to help evaluate organ and tissue functions.

SUMMARY:
This research study is studying a positron emission tomography (PET) agent called 18F-fluciclovine to evaluate how well 18F-fluciclovine-PET scans determine the extent of advanced prostate cancer that either has low prostate-specific membrane antigen (PSMA) expression or has neuroendocrine features.

The name of the study interventions are:

* 18F-fluciclovine-PET/CT scan
* Two research blood collections

DETAILED DESCRIPTION:
This research study is a pilot study, which is the first-time investigators are examining this study imaging agent, 18F-fluciclovine, for use in PSMA-low castration resistant and neuroendocrine prostate cancer detection.

18F-fluciclovine is approved by the U.S. Food and Drug Administration (FDA). It is approved for imaging the early stages of prostate cancer. It is not approved for imaging PSMA-low castration resistant or neuroendocrine prostate cancer. 18F-fluciclovine is a radiotracer for PET imaging that targets amino-acid receptors. Some information shows that both PSMA-low and neuroendocrine prostate tumors use amino acids for energy. The purpose of this study to determine if PSMA-low and neuroendocrine prostate cancer can be seen with 18F-fluciclovine-PET/CT. Secondary aims are better understanding of the role of amino acids and PSMA in PSMA low and neuroendocrine prostate cancer and how imaging tests can be used together to optimize treatments for PSMA-low and neuroendocrine prostate cancer.

Participants will receive a PSMA-PET/CT as part standard of care and as part of the study receive 18F-fluciclovine-PET/CT scan along with two research blood collections.

Blue Earth Diagnostics Inc. is supporting this research study by providing the 18Ffluciclovine and funding for the research study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed prostate cancer that is metastatic and one of the following: CRPC with PSMA-low disease defined by whole-body SUVmean ≤ 10 determined by standard-of-care 68Ga-PSMA-11 PET/CT imaging with at least 5 metastatic lesions OR NEPC pathology based on tumor biopsy. This may include morphology consistent with small cell carcinoma or mixed adenocarcinoma/NE features and/or IHC staining for NE markers. Participants should have at least 5 metastatic lesions.
* Must have either already had standard of care 68Ga-PSMA PET/CT scan or be planned for 68Ga-PSMA PET/CT scan before or after the planned 18F-fluciclovine-PET/CT.
* Age ≥18 years. Since no dosing or adverse event data are currently available on the use of 18F-fluciclovine in participants <18 years of age, and most prostate cancer occurs in the adult population, children are excluded from this study but will be eligible for future pediatric trials.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Ability and willingness to comply with the study procedures.
* The effects of 18F-fluciclovine on the developing human fetus are unknown. For this reason and because radiopharmaceuticals may be teratogenic, men must agree to use adequate contraception (barrier method of birth control; abstinence) prior to study entry and for 24 hours after the PET/CT scan is completed.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants with other known malignancy requiring treatment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 18F-fluciclovine.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Contraindications for PET/CT including:

  * Severe claustrophobia
* Any past or current condition that in the opinion of the study investigators would confound the results of the study or pose additional risk to the patient by their participation in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Fluciclovine and PSMA Uptake in PSMA Positive Tumors | Up to 6 months
  Number of 18F-fluciclovine positive lesions in PSMA-positive tumors on PET
  Number of fluciclovine positive tumors that are PSMA-negative
Fluciclovine and PSMA Uptake in PSMA Negative Tumors | up to 6 months
  Number of 18F-fluciclovine positive lesions in PSMA-negative tumors on PET

CONTACTS AND LOCATIONS:
Overall Officials: Heather Jacene, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Brigham and Womens Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu